CLINICAL TRIAL: NCT05978817
Title: Clinical Effectiveness of Damon Ultima Vs Conventional Brackets (A Randomized Clinical Trial)
Brief Title: Clinical Effectiveness of Damon Ultima Vs Conventional Brackets Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Nawar Ahmed Abed, Dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Damon Ultima brack treatment
Record Dates: First submitted 2023-04-16; First posted 2023-08-07 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Skeletal and Dental CL I Malocclusion Moderate Crowding

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Double (open label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Damon Ultima brackets (Experimental): Damon Ultima brackets
  Interventions: Device: Damon Ultima bracket
- conventional Roth appliance (Experimental): conventional Roth appliance
  Interventions: Device: Damon Ultima bracket

INTERVENTIONS:
Device: Damon Ultima bracket — It is metal twin bracket with their recommended arch wire
  Other Names: conventional Roth appliance

SUMMARY:
Compare the clinical performance, root resorption and pain perception between passive self-ligating Damon Ultema vs conventional brackets.

DETAILED DESCRIPTION:
Damon Ultima System was introduced and claimed to be the first true full expression orthodontic system designed for faster and more precise finishing. The brackets were completely reengineered to virtually eliminate play for precise control of rotation, angulation and torque. Moreover, the system used specially designed archwires regarding wire dimensions and shape to fulfill the manufacturers claim.

ELIGIBILITY:
Inclusion Criteria:

* 15-35 years of age patients who are healthy and without medications such as non-steroidal anti-inflammatory analgesics.
* Patients with Class I normal occlusion with moderate dental irregularity (with 4-6 irregularity index) requiring non-extraction treatment.
* Presence of all the permanent teeth apart from the third molars.
* Patients with good oral hygiene and periodontal health.
* Without previous orthodontic treatment/ functional appliances

Exclusion Criteria:

Patients will be excluded from recruitment if he had sever skeletal discrepancy that requires orthognathic surgery.

• Patients who have cleft lip or palate, hypodontia, or hyperdontia

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Occlusal outcomes assessment | 1 year
  1. Alignment, 2. Marginal ridge height, 3. Buccolingual inclination, 4. Overjet, 5. Occlusal contacts, 6. Occlusal relationships, 7. Interproximal contacts (1-7) Component: scores < 0.5 = 0. 0.5 to 1 mm =1. > 1 mm = 2. 8. Root angulation: Root parallelism = 0. Roots are not parallel = 1. Contacting adjacent tooth = 2. High scores on individual segments, or combinations of individual segments, may cause a case to become Incomplete.
  SO:
  the minimum value = 0 the maximum value = 16 the high score means = worse outcome the low score means = better outcome
Little Irregularity index: | 6 months
  This technique involves measuring the linear distance from anatomic contact point to the adjacent anatomic contact point of the mandibular anterior teeth , used to assess the changes in dental alignment throughout the study.
  initial irregularity index is (3 mm to 7mm) = worse out come and the final irregularity index is zero mm= best out come
Arch parameter measurement: | 1 year
  Arch length, arch width will be measured in millimeters and shape will be assessed by change from narrow shape arch to wide shape arch
Root alingment | 1 year
  Root movement in 3 plane of space will be evaluated at the end of the alignment phase after insertion of stainless steel wire which may will Tacke about 6 months and at the end of the treatment after about 6 months using CBCT. The inclination of upper and lower teeth will be assessed
Root resorption | 1 year
  Orthodontically induced inflammatory root resorption OIIRR will be assessed and the prevalence of root resorption will be calculated using CBCT radiographs.

SECONDARY OUTCOMES:
Patient experience and satisfaction | 1 year
  The pain perception will be assessed using visual analog scale (VAS) immediately after wire insertion, at 4, 24 hours, 3 days, 7 days, and immediately after each monthly visit (0 no pain, 3 simple pain, 100 very sever pain).
  Pain sensitivity questionnaire (PSQ) will be used to assess the patient reliability to pain. This will be done using the Arabic version of PSQ (The patient answer no or yes)

CONTACTS AND LOCATIONS:
Overall Officials: Dheaa H Al-Groosh, PHD, Principal Investigator — University of Baghdad
Locations (1):
- Nawar A jebory, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
randomized clinical trial